CLINICAL TRIAL: NCT04471220
Title: Examination of Exercise Capacity Under Various Oxygen Concentrations and Oxygen Flow Rates Using High Flow Nasal Cannula
Brief Title: Exercise Capacity Under Various FiO2 and Oxygen Flow Rates Using HFNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Hospital Organization Minami Kyoto Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2019-23
Record Dates: First submitted 2020-07-07; First posted 2020-07-15 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: High-flow Nasal Cannula; Exercise Capacity; Respiratory Failure
Keywords: HFNC; 6MWD
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low FIO2 and low flow rate under HFNC (Active Comparator): In this condition, patients have undergone 6MWT under the HFNC (FIO2 value that the minimum SpO2 value in a 6MWT is 86-88%, and a flow of 10 L/min).
  Interventions: Device: High-flow nasal cannula
- Low FIO2 and high flow rate under HFNC (Active Comparator): In this condition, patients have undergone 6MWT under the HFNC (FIO2 value that the minimum SpO2 value in a 6MWT is 86-88%, and a flow of 40-50 L/min).
  Interventions: Device: High-flow nasal cannula
- High FIO2 and low flow rate under HFNC (Active Comparator): In this condition, patients have undergone 6MWT under the HFNC (FIO2 value that the minimum SpO2 value in a 6MWT is 92-94%, and a flow of 10 L/min).
  Interventions: Device: High-flow nasal cannula
- High FIO2 and high flow rate under HFNC (Active Comparator): In this condition, patients have undergone 6MWT under the HFNC (FIO2 value that the minimum SpO2 value in a 6MWT is 92-94%, and a flow of 40-50 L/min).
  Interventions: Device: High-flow nasal cannula

INTERVENTIONS:
Device: High-flow nasal cannula — The nasal high flow therapy has enabled high flow oxygen to be derived through nasal cannula. This mode not only allows constant FiO2 during peak inspiratory flow but also confers benefits including a low level of continuous positive airway pressure with increased end-expiratory lung volume and reduced work of breathing, partly through intrinsic positive end-expiration pressure compensation and dead space washout. The inspired gases are warmed and humidified, improving comfort and possibly reducing airway inflammation, leading to improved drainage of respiratory secretions.

SUMMARY:
The purpose of this study is to compare the exercise capacity (6-min walking distance) under the following 4 conditions using High-flow nasal cannula (HFNC); 1. FIO2 value that the minimum SpO2 value in a 6-minute walking test (6MWT) is 86-88%, and a flow of 10 L/min 2. FIO2 value that the minimum SpO2 value in a 6MWT is 86-88%, and a flow of 40-50 L/min 3. FIO2 value that the minimum SpO2 value in a 6MWT is 92-94%, and a flow of 10 L/min 4. FIO2 value that the minimum SpO2 value in a 6MWT is 92-94%, and a flow of 40-50 L/min

DETAILED DESCRIPTION:
In the pervious study, the investigators demonstrated that 4 weeks of training using both high FIO2 and high flow through an HFNC significantly improved the 6MWD compared with training using a 6 L/min nasal cannula. However, it was unclear whether the effects of pulmonary rehabilitation under HFNC were due to high FIO2, high flow rate, or a synergistic effect. It is also unknown whether there are differences in the effects of pulmonary rehabilitation under HFNC for each underlying disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a minimum SPO2 of 88% or less during performing 6MWT under HFNC (FIO2 0.21 and a flow rate of 10L/min)
* Subjects who have been clinically stable for the last 2 weeks
* Subjects with written informed consent to participate in this study

Exclusion Criteria:

* Subjects with severe cardiovascular disease, liver disease, neurological disease, and renal failure
* Subjects who needed antimicrobial agent or steroid administration for pneumonia and exacerbation of respiratory disease in the last 2 weeks
* Subjects who cannot undergo 6MWT due to severe heart failure, arteriosclerosis obliterans or spinal disease

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-09-29 (Actual)

PRIMARY OUTCOMES:
Difference in 6MWD between two conditions ("Low FIO2 and high flow rate" and "High FIO2 and high flow rate") | through study completion, an average of 2 weeks

SECONDARY OUTCOMES:
Difference in 6MWD between four conditions | through study completion, an average of 2 weeks
Difference in SpO2 value during 6MWT between four conditions | through study completion, an average of 2 weeks
Difference in Pulse rate value during 6MWT between four conditions | through study completion, an average of 2 weeks
Difference in Dyspnea during 6MWT between four conditions | through study completion, an average of 2 weeks
Difference in lower limb fatigue during 6MWT between four conditions | through study completion, an average of 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- National Hospital Organization Minami Kyoto Hospital, Jōyō, Kyoto, Japan